CLINICAL TRIAL: NCT06215612
Title: ctDNA and MR Imaging Parameters as Possible Biomarkers in Primary Radiochemotherapy of Head and Neck Squamous Cell Carcinomas
Brief Title: ctDNA and MRI Parameters in Head and Neck Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Franziska Eckert (Other)
Responsible Party: Sponsor-Investigator, Franziska Eckert, Deputy Head of Department, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1452/2023
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood draw, MRI — Blood draw, MRI

SUMMARY:
Patients undergoing primary radiochhemotherapy for locally advanced head and neck squamous cell carcinomas are included in this study. In addition to standard of care treatment patients will undergo addiational blood draws and MR imaging studies. Circulating cell free tumor DNA will be analysed in the blood samples. BIological data, imaging data and clinical data (such as patient and tumor characteristics, oncologic outcome, side effects) will be analysed in a biomathematical modelling approach.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma head and neck
* Planned primary platinum based radiochemotherapy
* ECOG 0-2

Exclusion Criteria:

* Palliative therapy intent
* Not MR eligible

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with 50% decrease in ctDNA | 7 weeks after start of radiotherapy

SECONDARY OUTCOMES:
Completion of all planned MR imagings and blood tests | through study completion, an average of 7 weeks
Decrease of tumor volume | 7 weeks after start of radiotherapy

IPD SHARING:
Plan to Share IPD: No